CLINICAL TRIAL: NCT01423435
Title: A Pharmacokinetic Study of TRK-100STP -A Single Oral Administration Study in Japanese, Chinese, and South Korean Non-elderly Healthy Adult Males -
Brief Title: Study to Compare Pharmacokinetic Profiles of TRK-100STP in Japanese, Chinese, and South Korean Non-elderly Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 533-CL-006
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Adult Male; Pharmacokinetics of TRK-100-STP
Keywords: TRK-100STP; PK; beraprost sodium
MeSH Terms: interventions — beraprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Japanese (Experimental)
  Interventions: Drug: TRK-100STP
- Chinese (Experimental)
  Interventions: Drug: TRK-100STP
- South Korean (Experimental)
  Interventions: Drug: TRK-100STP

INTERVENTIONS:
Drug: TRK-100STP — oral
  Other Names: beraprost; Careload LA; YM533

SUMMARY:
A study to evaluate the pharmacokinetics and safety of TRK-100STP in Japanese, Chinese, and South Korean non-elderly healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: =<50.0 to 80.0> kg
* BMI: =<17.6 to 26.4>
* Subjects whose condition an investigator/subinvestigator has confirmed to be healthy by the date of drug administration, based on the screening test results

Exclusion Criteria:

* Subjects who received an investigational drug within 120 days prior to the screening test in other clinical trials or post-marketing studies
* Subjects who had 400 mL whole blood drawing within 90 days prior to the screening test, who had 200 mL whole blood drawing within 30 days prior to the screening test, or had component blood drawing within 14 days prior to the screening test
* Subjects who has received or will receive any drug treatment including over the counter (OTC) drugs within 7 days prior to the day of confinement
* Subjects whose vital signs are out of the standard level in one of the following parameters at the time of the screening test or the day of confinement: blood pressure, pulse rate, body temperature, and 12-lead ECG
* Subjects who have had upper Gastro-Intestinal (GI) symptoms within 7 days prior to the day of confinement (1 day prior to the drug administration): nausea, vomiting, or stomachache
* Subjects who have complications or history of liver diseases: viral hepatitis or chronic bronchitis
* Subjects who have complications or history of Cardio Vascular (CV) diseases: chronic heart failure, angina, or arrythmia that needs treatment
* Subjects who have complications or history of respiratory diseases: severe bronchial asthma or chronic bronchitis. History of pediatric asthma is not included
* Subjects who have complications or history of respiratory diseases: severe peptic ulceration or gastro-esophageal reflux disease. History of appendicitis is not included
* Subjects who have complications or history of renal diseases: acute renal failure, glomerulonephritis, or interstitial nephritis. History of calculus is not included
* Subjects who have complications or history of cerebrovascular diseases including cerebral infarction
* Subjects who have complications or history of malignant tumors
* Subjects in whom the daily amount of alcohol or smoking is excessive
* Subjects who have received beraprost

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic parameters of TRK-100STP such as maximum observed concentration (Cmax), area under the serum concentration-time curve (AUC) and terminal half-life (t1/2) | Up to 48 hours

SECONDARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, 12-lead electrocardiograms (ECGs) and lab tests | Up to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan